CLINICAL TRIAL: NCT03993314
Title: Comparing 1% Spinal Chloroprocaine to Low-dose Bupivacaine Using the Epidural Volume Extension Technique for Post-Partum Tubal Ligation
Brief Title: Optimizing Anesthesia for Post Partum Tubal Ligations
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment due to COVID-19 pandemic; chloroprocaine shortage
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mark Powell, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-300003361
Record Dates: First submitted 2019-06-17; First posted 2019-06-20 (Actual); Results first posted 2021-12-17 (Actual); Last update posted 2021-12-17 (Actual); Status verified 2021-12

CONDITIONS: Pregnancy Related
MeSH Terms: interventions — chloroprocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Bupivacaine (Active Comparator): 1 ml 0.5% isobaric bupivacaine (5 mg) + 15 mcg fentanyl intrathecal plus epidural volume extension (EVE)
  Interventions: Drug: Bupivacaine
- Chloroprocaine (Experimental): 5 ml 1% spinal chloroprocaine (50 mg) intrathecal plus epidural volume extension (EVE)
  Interventions: Drug: Chloroprocaine

INTERVENTIONS:
Drug: Chloroprocaine — Adding 5 cc 1% Chloroprocaine with 10 cc sterile saline in the epidural
  Arms: Chloroprocaine
Drug: Bupivacaine — 1 cc of 0.5% bupivacaine with 15 mcg fentanyl 10 cc of sterile saline in the epidural
  Arms: Bupivacaine

SUMMARY:
In this study, the investigators will compare CLOROTEKAL® (1% spinal chloroprocaine) to low-dose isobaric bupivacaine using the epidural volume extension (EVE) technique in patients undergoing post-partum tubal ligation (PPBTL). This will be a randomized, double-blinded study. Patients scheduled for PPBTL at the Women and Infants Center (WIC) will be eligible for enrollment in this study. Outcomes measured will include: ability to achieve an adequate level required for surgery (T6), rate of epidural activation, and duration of the block. The investigators hope to determine the usefulness of each drug using the EVE technique in the setting of PPBTL.

ELIGIBILITY:
Inclusion Criteria:

* Any patient scheduled for a postpartum tubal ligation at the Women and Infants Center will be eligible for the study

Exclusion Criteria:

* age less than 18 years old
* allergy to either local anesthetic class (amide or ester)
* contraindication to spinal anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-08-13 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2020-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark F Powell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bupivacaine | Chloroprocaine
Started | 9 | 6
Completed | 9 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine | Chloroprocaine | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.2 (4.5) | 27.0 (3.7) | 28.3 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.0 (7.1) | 31.7 (5.3) | 32.5 (6.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve a Level of Numbness of T6 or Higher
Description: Degree of analgesia is determined by the level of the block. Block level may be T1 (highest level of numbness), T2, T3, T4, T5, T6, T7,T8, T9 , T10, T11, T12, L1, L2, L3, or L4 (lowest level or numbness).
  A level of numbness of T6 or higher is required for an adequate surgical block. Participants are classified as having either an adequate level of numbness (T1, T2, T3, T4, T5, or T6) or an inadequate level (T7,T8, T9 , T10, T11, T12, L1, L2, L3, or L4).
Time Frame: 10 minutes after spinal injection
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
Participants
  Adequate level of numbness | 8 | 5
  Inadequate level of numbness | 1 | 1
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; Exact Farrington-Manning (Score) test of the null hypothesis that there is no difference between the proportion of patients achieving a level of numbness of T6 or higher between the two groups; Test type: Superiority; p = 0.757, Farrington-Manning (Score) test — Two-sided p-value

2. Primary Outcome: Level of Numbness
Description: The degree to which participants experience analgesia. Degree of analgesia is determined by the level of the block. Block level may be T1 (highest level of numbness), T2, T3, T4, T5, T6, T7,T8, T9 , T10, T11, T12, L1, L2, L3, or L4 (lowest level or numbness).
  Participants are assigned a numerical score according to level of the block. Numerical scores were assigned so that a higher score indicates better outcome (i.e., greater level of numbness):
  T1 = 16 points; T2 = 15 points; T3 = 14 points; T4 = 13 points; T5 = 12 points; T6 = 11 points; T7 = 10 points; T8 = 9 points; T9 = 8 points; T10 = 7 points; T11 = 6 points; T12 = 5 points; L1 = 4 points; L2 = 3 points; L3 = 2 points; L4 = 1 point
Time Frame: 10 minutes after spinal injection
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
score on a scale | 15 [13 to 16] | 12.5 [12 to 15]
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; Exact Wilcoxon test of the null hypothesis that there is no difference between the median level of numbness between the two groups; Test type: Superiority; p = 0.186, Wilcoxon (Mann-Whitney) — Two-sided p-value; Test performed was an exact test; no continuity correction was used

3. Secondary Outcome: Epidural Activation
Description: Number of patients who required epidural activation
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
Participants
  Epidural activated | 5 | 1
  Epidural not activated | 4 | 5
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; Exact Farrington-Manning (Score) test of the null hypothesis that there is no difference between the proportion of patients requiring epidural activation between the two groups; Test type: Superiority; p = 0.132, Farrington-Manning (Score) test — Two-sided p-value

4. Secondary Outcome: Supplemental Intravenous Sedation or General Anesthesia
Description: Number of patients who required supplemental intravenous sedation or general anesthesia
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
Participants
  Supplemental IV sedation or general anesthesia | 5 | 3
  No supplemental IV sedation or general anesthesia | 4 | 3
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; Exact Farrington-Manning (Score) test of the null hypothesis that there is no difference between the proportion of patients requiring supplemental IV sedation or general anesthesia between the two groups; Test type: Superiority; p = 0.833, Farrington-Manning (Score) test — Two-sided p-value

5. Secondary Outcome: Modified Bromage Score at 10 Minutes Post-injection
Description: The modified Bromage score is an ordinal scale ranging from 0 to 4 with higher values indicating greater levels of numbness.
  0 = ability to maintain leg lift for prolonged period; 1 = ability to lift legs briefly; 2 = ability to bend knees; 3 = ability to wiggle toes; 4 = no movement of lower extremities
Time Frame: 10 minutes after spinal injection
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
Participants
  0 = Ability to maintain leg lift for prolonged period | 1 | 0
  1 = Ability to lift legs briefly | 2 | 0
  2 = Ability to bend knees | 4 | 0
  3 = Ability to wiggle toes | 2 | 3
  4 = No movement of lower extremities | 0 | 3
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; Exact Wilcoxon test of the null hypothesis that there is no difference between the median modified Bromage score between the two groups; Test type: Superiority; p = 0.004, Wilcoxon (Mann-Whitney) — Two-sided p-value; Test performed was an exact test; no continuity correction was used

6. Secondary Outcome: Modified Bromage Score 60 Minutes After Intrathecal Injection
Description: as for outcome 5
Time Frame: 60 minutes after spinal injection
Measure: Count of Participants; unit: Participants
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
Participants
  0 = Ability to maintain leg lift for prolonged period | 2 | 0
  1 = Ability to lift legs briefly | 2 | 1
  2 = Ability to bend knees | 1 | 3
  3 = Ability to wiggle toes | 2 | 1
  4 = No movement of lower extremities | 2 | 1
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.674, Wilcoxon (Mann-Whitney) — Two-sided p-value; Test performed was an exact test; no continuity correction was used

7. Secondary Outcome: Time to PACU Discharge
Description: Time required for readiness for discharge from Post Anesthesia Care Unit (PACU)
Time Frame: Day of surgery
Measure: Median (Full Range); unit: minutes
Arm/Group | Bupivacaine | Chloroprocaine
Number analyzed (Participants) | 9 | 6
minutes | 57 [15 to 143] | 45 [21 to 93]
Statistical Analysis 1: Comparison: Bupivacaine vs Chloroprocaine; Log-rank test of the null hypothesis that there is no difference in the time to discharge from the Post Anesthesia Care Unit (PACU) between the two groups; Test type: Superiority; p = 0.196, Log Rank

ADVERSE EVENTS:
Time Frame: 1 day. Adverse event data were collected on day of post-partum tubal litigation (PPTL), from preoperative period to discharge from post anesthesia care unit (PACU).
Arm/Group | Bupivacaine | Chloroprocaine
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/14/NCT03993314/Prot_SAP_000.pdf